CLINICAL TRIAL: NCT04593810
Title: Effect of Automated Closed-Loop Ventilation Versus Conventional Ventilation on Duration and Quality of Ventilation ('ACTiVE') - a Randomized Clinical Trial in Intensive Care Unit Patients
Brief Title: Effect of Automated Closed-Loop Ventilation Versus Conventional Ventilation on Duration and Quality of Ventilation
Acronym: ACTiVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Marcus J. Schultz (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Catharina Ziekenhuis Eindhoven (Other); Reinier de Graaf Groep (Other); Flevoziekenhuis (Other); Leiden University Medical Center (Other); Canisius-Wilhelmina Hospital (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Diakonessenhuis, Utrecht (Other); Ospedale Policlinico San Martino (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr. Marcus J. Schultz, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTiVE
Record Dates: First submitted 2020-10-11; First posted 2020-10-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Ventilator-free Days; Quality of Breathing
Keywords: Automated invasive ventilation; Closed-loop invasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTELLiVENT-ASV (Experimental): Use of INTELLIVENT-ASV after intubation and during all mechanical ventilation in the ICU.
  Interventions: Procedure: INTELLiVENT-ASV
- Conventional ventilation (Active Comparator): Use of conventional ventilation after intubation and during all mechanical ventilation in the ICU.
  Interventions: Procedure: CONVENTIONAL VENTILATION

INTERVENTIONS:
Procedure: INTELLiVENT-ASV — INTELLiVENT-ASV is activated as soon possible. The sensors for ETCO2 and SpO2 are connected and activated. Patient's gender and height are set on the ventilator and patient condition is chosen if applicable.
  Arms: INTELLiVENT-ASV
Procedure: CONVENTIONAL VENTILATION — Conventional ventilation consists of VCV or PCV and PSV, depending on patient's activity. None of the semi or fully automated modes of ventilation is allowed at any time.
  Arms: Conventional ventilation

SUMMARY:
INTELLiVENT-Adaptive Support Ventilation (ASV) is a fully automated closed-loop mode of mechanical ventilation available on commercial ventilators. Evidence for clinical benefit of INTELLiVENT-ASV in comparison to non-automated ventilation is lacking.

The ACTiVE study is an international, multicenter, randomized controlled trial in invasively ventilated ICU patients with the objective to compare INTELLiVENT-ASV to conventional ventilation. We hypothesise that INTELLiVENT-ASV shortens the duration of ventilation. The secondary hypothesis is that INTELLiVENT-ASV improves the quality of breathing.

DETAILED DESCRIPTION:
Objective

The primary objective of this trial is to compare INTELLiVENT-ASV with non-automated ventilation in critically ill intensive care unit (ICU) patients with respect to ventilation duration. One secondary aim is to test whether INTELLiVENT-ASV improves quality of breathing, expressed as the proportion of breath within lung-protective margins, in a time frame of 24 hours early after start of invasive ventilation.

Study design

International, multicenter, superiority randomized clinical trial in critically ill, intubated and ventilated adult ICU patients with an anticipated duration of ventilation of at least 24 hours.

Study population

Adult patients admitted to ICUs in the Netherlands and Italy.

Sample size calculation

The sample size is based on the hypothesis that INTELLiVENT-ASV will shorten ventilation duration by 1.5 days with no changes in mortality rate. Based on previously performed studies a sample of 1,200 patients (600 in each treatment group) is needed to have beta of 80% power and a two-tailed alpha of 0.05, to detect a mean between-group difference of 1.5 VFD-28, allowing a dropout rate of 5%. By including 1,200 patients, this study will be sufficiently powered to detect differences in the secondary endpoint, which is quality of breathing.

Methods:

Within one hour of start of ventilation in the ICU, patients are randomly assigned in a 1:1 ratio to INTELLiVENT-ASV or non-automated ventilation. Randomization will be stratified by center. As soon as possible after randomization, but within a maximum of 72 hours, deferred consent is obtained from the legal representative of the patient.

INTELLiVENT-ASV In patients who are randomized to INTELLiVENT-ASV, the ventilator is switched to this fully automated mode as soon possible. The sensors for end-tidal carbon dioxide (ETCO2) and pulse oximetry (SpO2) are connected and activated in the ventilator. Patient's gender and height are set on the ventilator and patient condition is chosen if applicable. If needed, the targets zones for ETCO2 and SpO2 are adjusted. The default alarm limits are accepted.

It is advised to enable QuickWean in all patients. The use of the automated Spontaneous Breathing Trial (SBT) function is left to the discretion of the clinician.

CONVENTIONAL VENTILATION Patients who are randomized to conventional ventilation will be ventilated with a mode that is not fully automated, thus standard volume controlled (VCV) or pressure controlled ventilation (PCV), and pressure support ventilation (PSV), depending on patient's activity. None of the following semi or fully automated modes of ventilation is allowed at any time: Neurally Adjusted Ventilatory Assist (NAVA), SmartCare/PS, Proportional Assist Ventilation (PAV), or the predecessor of INTELLiVENT-ASV named ASV.

In all patients who receive assist ventilation (i.e., VCV or PCV), three times a day it should be checked whether the patient can accept supported ventilation (i.e., PSV); this should also be tried when the patient shows respiratory muscle activity during assist ventilation, or in case of patient-ventilator asynchrony.

Patients can be subjected to SBTs using either a T-piece or ventilation with minimal support (pressure support level < 10 cm H2O). An SBT is deemed successful when the following criteria are met for at least 30 minutes, i.e., respiratory rate < 35/min, peripheral oxygen saturation > 90%, increase < 20% of heart rate and blood pressure, and no signs of anxiety and diaphoresis.

In both groups patients are extubated if standard extubation criteria are fulfilled, i.e., normal body temperature, patient awake and responsive/cooperative, adequate cough reflex, adequate oxygenation, hemodynamically stable, and adequate lung function.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the participating ICUs
* intubated and receiving invasive ventilation
* anticipated duration of ventilation of at least 24 hours

Exclusion Criteria:

* age below 18 years
* patients with suspected or confirmed pregnancy
* invasive ventilation > 1 hour in the ICU
* invasive ventilation > 6 hours directly preceding the current ICU admission
* participation in another interventional trial using similar endpoints
* after recent pneumectomy or lobectomy
* morbid obesity (body mass index > 40 kg/m2)
* premorbid restrictive pulmonary disease
* unreliable pulse oximetry (secondary to carbon monoxide poisoning or sickle cell disease)
* any neurologic diagnosis that can prolong duration of mechanical ventilation, e.g., Guillain-Barré syndrome, high spinal cord lesion or amyotrophic lateral sclerosis, multiple sclerosis, or myasthenia gravis
* patients receiving or planned to receive veno-venous, veno-arterial or arterio-venous extracorporeal membrane oxygenation (ECMO)
* unavailability of INTELLiVENT-ASV (no ventilator available with this ventilation mode)
* previously randomized in this study
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days and alive at day 28 | first 28 days after start of ventilation
  The number of days from day 1 to day 28 the patient is alive and breathes without assistance of the mechanical ventilator, if the period of unassisted breathing lasted at least 24 consecutive hours

SECONDARY OUTCOMES:
Quality of breathing | 24 hours early after start of invasive ventilation.
  Proportion of breaths within lung-protective margins
Duration of ventilation | first 28 days after start of ventilation
  Duration of ventilation in survivors
Length of stay | first 90 days after start of ventilation
  Length of stay in the intensive care unit and in the hospital
Mortality | first 90 days after start of ventilation
  Any death during ICU- or hospital-stay, at day 28 and day 90
Pulmonary complications | daily until ICU discharge or day 28
  Development of ARDS, severe hypoxemia, severe hypercapnia, severe atelectasis, pneumothorax and ventilator-associated pneumonia
Rescue therapies for severe hypoxemia or severe atelectasis | daily until ICU discharge or day 28
  Incidence of use of rescue therapies for severe hypoxemia or severe atelectasis: recruitment maneuver, prone positioning, bronchoscopy for opening atelectasis
Extubation failure | daily until ICU discharge or day 28
  Extubation with need for reintubation within 24 hours
Maximal inspiratory pressure (MIP) | within 24 hours after extubation
  Maximal inspiratory pressure measured after extubation at centers that can collect this data
Quality of Life questionnaire | day 28 after start of ventilation
  The European Quality of life 5 Dimensions 5 Levels questionnaire (EQ-5D-5L) is used to assess health-related quality of life status in adults. It consists of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels (from 1 to 5) that are described by statements appropriate to that dimension. Higher values mean worse quality of life. The evaluation includes a visual analogue scale to quantitative measure the overall health status. This scale has a range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Janneke Horn, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center; Frederique Paulus, PhD, Study Director — Department of Intensive Care, Academic Medical Center; Marcus J Schultz, MD,PhD, Study Director — Department of Intensive Care, Academic Medical Center
Locations (10):
- Italy (2):
  - Ospedale Policlinico San Martino, Genoa
  - Policlinico San Matteo Fondazione IRCCS, Pavia
- Netherlands (8):
  - Flevoziekenhuis, Almere Stad
  - Academic Medical Center, Intensive Care, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Leiden UMC, Leiden
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Diakonessenhuis, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sinnige JS, Buiteman-Kruizinga LA, Horn J, Paulus F, Schultz MJ, Serpa Neto A; ACTiVE Investigators and the Protective Ventilation Network. Effect of Automated Closed-Loop Ventilation vs Protocolized Conventional Ventilation on Ventilator-Free Days in Critically Ill Adults: A Randomized Clinical Trial. JAMA. 2025 Dec 8:e2524384. doi: 10.1001/jama.2025.24384. Online ahead of print. PMID 41361939
- [Derived] Botta M, Tsonas AM, Sinnige JS, De Bie AJR, Bindels AJGH, Ball L, Battaglini D, Brunetti I, Buiteman-Kruizinga LA, van der Heiden PLJ, de Jonge E, Mojoli F, Robba C, Schoe A, Paulus F, Pelosi P, Neto AS, Horn J, Schultz MJ; ACTiVE collaborative group. Effect of Automated Closed-loop ventilation versus convenTional VEntilation on duration and quality of ventilation in critically ill patients (ACTiVE) - study protocol of a randomized clinical trial. Trials. 2022 Apr 23;23(1):348. doi: 10.1186/s13063-022-06286-w. PMID 35461264

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04593810/SAP_002.pdf